CLINICAL TRIAL: NCT01137812
Title: A Randomized, Double-Blind, Active-Controlled, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Canagliflozin Versus Sitagliptin in the Treatment of Subjects With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin and Sulphonylurea Therapy
Brief Title: The CANTATA-D2 Trial (CANagliflozin Treatment And Trial Analysis - DPP-4 Inhibitor Second Comparator Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017185; 28431754DIA3015 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Results first posted 2013-05-17 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Canagliflozin; Sitagliptin (Januvia); Metformin; Sulphonylurea; Hemoglobin A1c; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Canagliflozin; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Canagliflozin 300 mg (Experimental): Each patient will receive 300 mg of canagliflozin once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea
  Interventions: Drug: Canagliflozin 300 mg; Drug: Metformin; Drug: Sulphonylurea
- Sitagliptin 100 mg (Active Comparator): Each patient will receive 100 mg of sitagliptin once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea
  Interventions: Drug: Sitagliptin 100 mg; Drug: Metformin; Drug: Sulphonylurea

INTERVENTIONS:
Drug: Sitagliptin 100 mg — One 100 mg capsule once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea
  Arms: Sitagliptin 100 mg
Drug: Canagliflozin 300 mg — One 300 mg capsule once daily for 52 weeks with protocol-specified doses of metformin and sulphonylurea
  Arms: Canagliflozin 300 mg
Drug: Metformin — Patients will continue to take background therapy with Metformin for T2DM at maximally or near-maximally effective protocol-specified doses for the duration of the study.
Drug: Sulphonylurea — Patients will continue to take background therapy with Sulphonylurea for T2DM at maximally or near-maximally effective protocol-specified doses for the duration of the study.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of canagliflozin compared with sitagliptin in patients with type 2 diabetes mellitus who are receiving treatment with metformin and sulphonylurea and have inadequate glycemic (blood sugar) control.

DETAILED DESCRIPTION:
Canagliflozin is a drug that is being tested to see if it may be useful in treating patients diagnosed with type 2 diabetes mellitus (T2DM). This is a randomized (study drug assigned by chance), double-blind (neither the patient or the study doctor will know the name of the assigned treatment), multicenter study to determine the efficacy, safety, and tolerability of canagliflozin 300 mg compared to sitagliptin 100 mg (an antihyperglycemic drug) in patients with T2DM who are not achieving an adequate response from current antihyperglycemic therapy with metformin and sulphonylurea to control their diabetes. Approximately 720 patients with T2DM who are receiving combination therapy with metformin and sulphonylurea will receive the addition of once-daily treatment with canagliflozin 300 mg or sitagliptin 100 mg capsules for 52 weeks. Patients will participate in the study for approximately 59 to 72 weeks. During treatment, patients will be monitored for safety by review of adverse events, results from laboratory tests, 12-lead electrocardiograms (ECGs), vital signs measurements, body weight, physical examinations, and self monitored blood glucose (SMBG) measurements. The primary outcome measure in the study is the effect of canagliflozin compared to sitagliptin on hemoglobin A1c (HbA1c) after 52 weeks of treatment. Study drug will be taken orally (by mouth) once daily before the first meal each day unless otherwise specified. Patients will take single-blind placebo for 2 weeks before randomization. After randomization, patients in the study will take double-blind canagliflozin 300 mg or matching sitagliptin 100 mg for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of T2DM and be currently treated with metformin and sulphonylurea
* Patients in the study must have a HbA1c between >=7 and <=10.5% and a fasting plasma glucose (FPG) <300 mg/dL (16.7 mmol/L)

Exclusion Criteria:

* History of diabetic ketoacidosis, type 1 diabetes mellitus (T1DM), pancreas or beta cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy
* or a severe hypoglycemic episode within 6 months before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2010-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (184):
- United States (85):
  - Mobile, Alabama
  - Goodyear, Arizona
  - Mesa, Arizona
  - Escondido, California
  - Fresno, California
  - Greenbrae, California
  - La Mesa, California
  - Laguna Hills, California
  - Lancaster, California
  - Long Beach, California
  - Los Angeles, California
  - Norwalk, California
  - Pismo Beach, California
  - Roseville, California
  - Spring Valley, California
  - Walnut Creek, California
  - Watsonville, California
  - Denver, Colorado
  - Northglenn, Colorado
  - Milford, Connecticut
  - Bradenton, Florida
  - Cape Coral, Florida
  - Clearwater, Florida
  - Delray Beach, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Lewiston, Idaho
  - Chicago, Illinois
  - O'Fallon, Illinois
  - Springfield, Illinois
  - Topeka, Kansas
  - Bowling Green, Kentucky
  - Lexington, Kentucky
  - Madisonville, Kentucky
  - Baton Rouge, Louisiana
  - Mandeville, Louisiana
  - Metairie, Louisiana
  - Sunset, Louisiana
  - Brockton, Massachusetts
  - Saint Clair Shores, Michigan
  - Southfield, Michigan
  - Dakota Dunes, Nebraska
  - Toms River, New Jersey
  - Albuquerque, New Mexico
  - West Seneca, New York
  - Calabash, North Carolina
  - Greensboro, North Carolina
  - Moerhead City, North Carolina
  - Morganton, North Carolina
  - Cincinnati, Ohio
  - Gallipolis, Ohio
  - Marion, Ohio
  - Mason, Ohio
  - Toledo, Ohio
  - Zanesville, Ohio
  - Beaver, Pennsylvania
  - Bensalem, Pennsylvania
  - Norristown, Pennsylvania
  - Perryopolis, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Pottstown, Pennsylvania
  - Greenville, South Carolina
  - Spartanburg, South Carolina
  - Johnson City, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Killeen, Texas
  - Richardson, Texas
  - San Antonio, Texas
  - Schertz, Texas
  - Sugar Land, Texas
  - Burke, Virginia
  - Danville, Virginia
  - Falls Church, Virginia
  - Hampton, Virginia
  - Henrico, Virginia
  - Manassas, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Selah, Washington
  - Tacoma, Washington
- Austria (2):
  - Salzburg
  - Vienna
- Belgium (2):
  - Hedersem (Aalst)
  - Tremelo
- Brazil (9):
  - Belém
  - Brasília
  - Fortaleza
  - Goiânia
  - Marília
  - Passo Fundo
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
- Canada (12):
  - Calgary, Alberta
  - Red Deer, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Brampton, Ontario
  - Oshawa, Ontario
  - Toronto, Ontario
  - Charlottetown, Prince Edward Island
  - Sherbrooke, Quebec
  - Ville, Laint-Laurent, Quebec
  - Pointe-Claire
  - Toronto
- Denmark (5):
  - Aalborg
  - Ballerup Municipality
  - Gentofte Municipality
  - Vejle
  - Vipperoed
- France (8):
  - Bondy
  - Dijon
  - Marseille
  - Nantes
  - Narbonne
  - Paris
  - Pessac
  - Saint-Etienne
- Germany (5):
  - Berlin
  - Dresden
  - Eisenach
  - Großheirath
  - Meißen
- India (7):
  - Bangalore
  - Coimbatore
  - Hyderabad
  - Jaipur
  - Nagpur
  - Nashik
  - Pune
- Israel (6):
  - Beersheba
  - Jerusalem
  - Kfar Saba
  - Nazareth
  - Rishon LeZiyyon
  - Tel Aviv
- Malaysia (4):
  - Ipoh
  - Johor Bahru
  - Kelantan
  - Kuala Selangor
- Netherlands (7):
  - Breda
  - Eindhoven
  - Groningen
  - Leiderdorp
  - Rotterdam
  - Velp Gld
  - Zoetermeer
- New Zealand (5):
  - Christchurch
  - Dunedin
  - Rotorua
  - Tauranga
  - Wellington
- Poland (11):
  - Bialystok
  - Chrzanów
  - Gdansk
  - Kamieniec Ząbkowicki
  - Krakow
  - Lublin
  - Sobótka
  - Sopot
  - Torun
  - Wroclaw
  - Zabrze
- Singapore, Singapore
- South Korea (5):
  - Busan
  - Daegu
  - Jeonju
  - Seongnam
  - Seoul
- Ukraine (10):
  - Dnipro
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Odesa
  - Poltava
  - Sumy
  - Ternopil
  - Vinnitsa
  - Zaporizhzhya

REFERENCES:
- [Derived] Cai J, Delahanty LM, Akapame S, Slee A, Traina S. Impact of Canagliflozin Treatment on Health-Related Quality of Life among People with Type 2 Diabetes Mellitus: A Pooled Analysis of Patient-Reported Outcomes from Randomized Controlled Trials. Patient. 2018 Jun;11(3):341-352. doi: 10.1007/s40271-017-0290-4. PMID 29313267
- [Derived] Qiu R, Balis D, Xie J, Davies MJ, Desai M, Meininger G. Longer-term safety and tolerability of canagliflozin in patients with type 2 diabetes: a pooled analysis. Curr Med Res Opin. 2017 Mar;33(3):553-562. doi: 10.1080/03007995.2016.1271780. Epub 2017 Jan 4. PMID 27977934
- [Derived] Schernthaner G, Lavalle-Gonzalez FJ, Davidson JA, Jodon H, Vijapurkar U, Qiu R, Canovatchel W. Canagliflozin provides greater attainment of both HbA1c and body weight reduction versus sitagliptin in patients with type 2 diabetes. Postgrad Med. 2016 Nov;128(8):725-730. doi: 10.1080/00325481.2016.1210988. Epub 2016 Jul 26. PMID 27391951
- [Derived] Watts NB, Bilezikian JP, Usiskin K, Edwards R, Desai M, Law G, Meininger G. Effects of Canagliflozin on Fracture Risk in Patients With Type 2 Diabetes Mellitus. J Clin Endocrinol Metab. 2016 Jan;101(1):157-66. doi: 10.1210/jc.2015-3167. Epub 2015 Nov 18. PMID 26580237
- [Derived] Lavalle-Gonzalez FJ, Eliaschewitz FG, Cerdas S, Chacon Mdel P, Tong C, Alba M. Efficacy and safety of canagliflozin in patients with type 2 diabetes mellitus from Latin America. Curr Med Res Opin. 2016;32(3):427-39. doi: 10.1185/03007995.2015.1121865. Epub 2016 Jan 14. PMID 26579834
- [Derived] Bailey RA, Vijapurkar U, Meininger G, Rupnow MF, Blonde L. Diabetes-Related Composite Quality End Point Attainment: Canagliflozin Versus Sitagliptin Based on a Pooled Analysis of 2 Clinical Trials. Clin Ther. 2015 May 1;37(5):1045-54. doi: 10.1016/j.clinthera.2015.02.020. Epub 2015 Mar 18. PMID 25795432
- [Derived] Polidori D, Mari A, Ferrannini E. Canagliflozin, a sodium glucose co-transporter 2 inhibitor, improves model-based indices of beta cell function in patients with type 2 diabetes. Diabetologia. 2014 May;57(5):891-901. doi: 10.1007/s00125-014-3196-x. Epub 2014 Mar 1. PMID 24585202
- [Derived] Schernthaner G, Gross JL, Rosenstock J, Guarisco M, Fu M, Yee J, Kawaguchi M, Canovatchel W, Meininger G. Canagliflozin compared with sitagliptin for patients with type 2 diabetes who do not have adequate glycemic control with metformin plus sulfonylurea: a 52-week randomized trial. Diabetes Care. 2013 Sep;36(9):2508-15. doi: 10.2337/dc12-2491. Epub 2013 Apr 5. PMID 23564919

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of canagliflozin compared with sitaglitin in patients with type 2 diabetes mellitus with inadequate control, despite treatment with metformin and sulphonylureas. The study was conducted between 30 June 2010 and 09 March 2012 and recruited patients from 140 study centers located in 17 countries worldwide.
Pre-assignment Details: A total of 756 patients were randomly allocated to the 2 treatment arms in the study. 755 patients received at least 1 dose of study drug and were included in the modified intent-to-treat (mITT) analysis set and the safety analysis set.
Groups:
- Canagliflozin 300 mg: Each patient received 300 mg of canagliflozin once a day for 52 weeks with protocol-specified doses of metformin and sulphonylurea.
- Sitagliptin 100 mg: Each patient received 100 mg of sitagliptin once a day for 52 weeks with protocol-specified doses of metformin and sulphonylurea.
Period: Overall Study
Arm/Group | Canagliflozin 300 mg | Sitagliptin 100 mg
Started | 377 | 378
Completed | 254 | 210
Not Completed | 123 | 168
Not completed — Adverse Event | 21 | 14
Not completed — Lost to Follow-up | 6 | 8
Not completed — Physician Decision | 25 | 17
Not completed — Protocol Violation | 5 | 4
Not completed — Withdrawal by Subject | 5 | 13
Not completed — Death | 2 | 0
Not completed — Patient met glycemic withdrawal criteria | 40 | 85
Not completed — Other | 19 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canagliflozin 300 mg | Sitagliptin 100 mg | Total
Number analyzed (Participants) | 377 | 378 | 755
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 304 | 307 | 611
  >=65 years | 73 | 71 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (9.62) | 56.6 (9.33) | 56.5 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 163 | 333
  Male | 207 | 215 | 422
Region Treated [Number; unit: participants]
  AUSTRIA | 4 | 2 | 6
  BELGIUM | 3 | 2 | 5
  BRAZIL | 76 | 80 | 156
  CANADA | 41 | 45 | 86
  DENMARK | 2 | 5 | 7
  FRANCE | 5 | 6 | 11
  GERMANY | 5 | 5 | 10
  INDIA | 33 | 23 | 56
  ISRAEL | 7 | 3 | 10
  MALAYSIA | 10 | 14 | 24
  NETHERLANDS | 2 | 1 | 3
  NEW ZEALAND | 11 | 13 | 24
  POLAND | 20 | 25 | 45
  SINGAPORE | 2 | 2 | 4
  SOUTH KOREA | 7 | 12 | 19
  UKRAINE | 27 | 19 | 46
  UNITED STATES | 122 | 121 | 243

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 52
Description: The table below shows the least-squares (LS) mean change in HbA1c from Baseline to Week 52 for each treatment group. The statistical analysis shows the treatment difference (ie, between canagliflozin and sitagliptin) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 52
Population: This analysis used the modified intent-to-treat analysis set (all patients who were randomly assigned to a treatment group and received at least 1 dose of study drug). The last-observation-carried-forward method was applied when the Week 52 values were missing. The table includes only patients with both baseline and post baseline values.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 374 | 365
Percent | -1.03 (0.048) | -0.66 (0.049)
Statistical Analysis 1: Comparison: Canagliflozin 300 mg vs Sitagliptin 100 mg; If the hypothesis of non-inferiority of canagliflozin to sitagliptin at Week 52 was demonstrated (ie, upper bound of the 95% Confidence Interval of the treatment difference [canagliflozin minus sitagliptin] was less than 0.3) and the upper bound was less than 0.0, the superiority of the canagliflozin dose relative to sitagliptin would be concluded; Test type: Non-Inferiority or Equivalence — Power calculation: assuming a difference between canagliflozin and sitagliptin of 0.0% and a common standard deviation of 1.0%, and using a 2-sample, 1-sided t-test with a Type I error rate of 0.025, it was estimated that 234 patients per group would provide approximately 90% power to demonstrate non-inferiority with the non-inferiority margin of 0.3, comparing canagliflozin with sitagliptin; p < 0.05, ANCOVA; Least-Squares Mean Difference = -0.37, 95% CI 2-sided [-0.500 to -0.250], Standard Error of Mean 0.064

2. Secondary Outcome: Percentage of Patients With HbA1c <7% at Week 52
Description: The table below shows the percentage of patients with HbA1c <7% at Week 52 in each treatment group. The statistical analysis shows the treatment difference (ie, between canagliflozin and sitagliptin) in the percentage.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 374 | 365
Percentage of patients | 47.6 | 35.3
Statistical Analysis 1: Comparison: Canagliflozin 300 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 1.80, 95% CI 2-sided [1.30 to 2.48]

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 52
Description: The table below shows the least-squares (LS) mean change in FPG from Baseline to Week 52 for each treatment group. The statistical analysis shows the treatment difference (ie, between canagliflozin and sitagliptin) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 373 | 365
mg/dL | -29.9 (2.201) | -5.85 (2.232)
Statistical Analysis 1: Comparison: Canagliflozin 300 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -24.1, 95% CI 2-sided [-29.89 to -18.24]

4. Secondary Outcome: Percent Change in Body Weight From Baseline to Week 52
Description: The table below shows the least-squares (LS) mean percent change in body weight from Baseline to Week 52 for each treatment group. The statistical analysis shows the treatment difference (ie, between canagliflozin and sitagliptin) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 375 | 367
Percent change | -2.5 (0.2) | 0.3 (0.2)
Statistical Analysis 1: Comparison: Canagliflozin 300 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.8, 95% CI 2-sided [-3.3 to -2.2], Standard Error of Mean 0.3

5. Secondary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline to Week 52
Description: The table below shows the least-squares (LS) mean change in SBP from Baseline to Week 52 for each treatment group. The statistical analysis shows the treatment difference (ie, between canagliflozin and sitagliptin) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 375 | 367
mmHg | -5.06 (0.656) | 0.85 (0.666)
Statistical Analysis 1: Comparison: Canagliflozin 300 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -5.91, 95% CI 2-sided [-7.642 to -4.175], Standard Error of Mean 0.883

6. Secondary Outcome: Percent Change in Triglycerides From Baseline to Week 52
Description: The table below shows the mean percent change in triglycerides from Baseline to Week 52 for each treatment group. The statistical analysis shows the treatment difference (ie, between canagliflozin and sitagliptin) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 365 | 353
Percent change | 9.6 (2.8) | 11.9 (2.9)
Statistical Analysis 1: Comparison: Canagliflozin 300 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.554, ANCOVA; Least-Squares Mean Difference = -2.3, 95% CI 2-sided [-9.8 to 5.3], Standard Error of Mean 3.9

7. Secondary Outcome: Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 52
Description: The table below shows the mean percent change in HDL-C from Baseline to Week 52 for each treatment group. The statistical analysis shows the treatment difference (ie, between canagliflozin and sitagliptin) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Canagliflozin 300 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 364 | 353
Percent change | 7.6 (0.9) | 0.6 (0.9)
Statistical Analysis 1: Comparison: Canagliflozin 300 mg vs Sitagliptin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = 7.0, 95% CI 2-sided [4.6 to 9.3], Standard Error of Mean 1.2

ADVERSE EVENTS:
Time Frame: Adverse events were reported for the duration of the study; each patient participated in the study for approximately 52 weeks.
Description: The total number of adverse events listed in the "Other (non-Serious) Adverse Events" table are based upon a cut-off of greater than or equal to 5 percent of patients experiencing the adverse event in any treatment arm.
Arm/Group | Canagliflozin 300 mg | Sitagliptin 100 mg
Serious Adverse Events (participants affected / at risk) | 24/377 | 21/378
Other Adverse Events (participants affected / at risk) | 157/377 | 159/378
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canagliflozin 300 mg (N=377) | Sitagliptin 100 mg (N=378)
Angina unstable (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Gallbladder oedema (Hepatobiliary disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Leptospirosis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cervical cord compression (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canagliflozin 300 mg (N=377) | Sitagliptin 100 mg (N=378)
Diarrhoea (Gastrointestinal disorders) | 17 | 26
Influenza (Infections and infestations) | 22 | 15
Nasopharyngitis (Infections and infestations) | 33 | 38
Upper respiratory tract infection (Infections and infestations) | 33 | 21
Urinary tract infection (Infections and infestations) | 15 | 19
Hypoglycaemia (Metabolism and nutrition disorders) | 66 | 75
Headache (Nervous system disorders) | 29 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.